CLINICAL TRIAL: NCT01393691
Title: Interventions for Nighttime Fears in Preschool Children: Assessment of Predictors and Outcomes
Brief Title: A Clinical Research Studying Interventions for Nighttime Fears in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: alan apter (Other)
Responsible Party: Sponsor-Investigator, alan apter, Director of psychological medicine department at Schneider; Professor at Sackler School of medicine, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6191
Record Dates: First submitted 2011-07-03; First posted 2011-07-13 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Nighttime Fears
Keywords: nighttime fears; anxiety; sleep; actigraphy; intervention
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT with parent combined play (Experimental): This is a CBT adaptation designed for preschool children, which includes multiple standard cognitive-behavioral techniques, namely psycho-education, problem solving via play, gradual exposure and reinforcement management.
  Interventions: Behavioral: CBT with parent involved play
- Triadic expressive play therapy (Active Comparator): Based on expressive play therapy guidelines, children and their parents will express themes concerning bedtime routines and fears via play.
  Interventions: Behavioral: Triadic expressive play therapy

INTERVENTIONS:
Behavioral: CBT with parent involved play — This is a CBT adaptation designed for preschool children, which includes multiple standard cognitive-behavioral techniques, namely psycho-education, problem solving via play, gradual exposure and reinforcement management.
  Arms: CBT with parent combined play
Behavioral: Triadic expressive play therapy — Based on expressive play therapy guidelines, children and their parents will express themes concerning bedtime routines and fears via play.
  Arms: Triadic expressive play therapy

SUMMARY:
Nighttime fears (NTF) and sleep disruptions in preschool children continue to be major problems in clinical services. The aim of this study is to test the efficacy of two interventions designed for preschool children suffering from NTF: (a) a CBT adaptation combining parent involved play, which will include multiple standard cognitive-behavioral techniques, namely psycho-education, problem solving via play, gradual exposure and reinforcement management; and (b) Triadic Expressive Play Therapy, based on Virginia Axline's (1947) eight basic principles of play therapy. Parents will take an active part both in and in between treatment sessions in both intervention groups. In addition to the review of the outcomes of these interventions, the proposed study aims to identify variables that moderate and mediate treatment effects.

In an attempt to meet these aims, the investigators will recruit 90 children suffering severe NTF and their parents who seek treatment. At baseline the investigators will assess children's NTF and general fears, sleep patterns and disruptions, behavior problems and potential moderators (i.e. playfulness, oppositionality, desire for control and parental anxiety). Assessment will be based on both objective and subjective measures, including interviews with the child and parents, questionnaires and actigraphy. The investigators will then randomly assign these children to one of two conditions: CBT with parent involved play or Triadic expressive play therapy. Possible mediators (i.e. the therapeutic alliance, patient compliance, motivation etc.) will be evaluated after each of the active intervention sessions. The effects of the interventions will be assessed by comparing four time points: baseline, first week of intervention, 1 month and 6 months subsequent to administration.

The main hypotheses of the proposed study are: (a) A positive correlation will be found between the severity of NTF and the severity of sleep disruption at baseline, and a reduction in NTF will be associated with an improvement in sleep; (b) Both interventions will significantly reduce nighttime fears, but greater impact will be evident in the CBT group; (c) Higher levels of playfulness and lower levels of oppositionality and desire for control, as well as parental anxiety will predict desirable outcomes. (d) Stronger therapeutic alliances, in addition to higher levels of motivation and compliance will be associated with greater intervention effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* NTF exist for a minimum of 2 months, with significant adverse impact on the child and the family, requiring parental involvement for at least two nights per week to comfort the child.

Exclusion Criteria:

* major health or neurological-developmental problems
* concurrent psychiatric treatment
* concurrent psychotherapy or any other intervention aimed at reducing the child's nighttime fears.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2011-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
nighttime fear and sleep logs | 1 week- 6 months
  Parents will be asked to report the level of their child's fear in the fear diary every night after bedtime, and every morning after the child has awoken from slumber. In addition, they will be asked to document the influence fears had on their child's sleep and bedtime routine, and the coping strategies that were implemented by themselves and by their child during the night.
Nighttime fears interview (child) and nighttime fears questionnaire (parents) | 1 week -6months
  Children will be interviewed regarding the content, frequency and severity of their nighttime fears. Parents will complete a questionnaire regarding these issues.

SECONDARY OUTCOMES:
Activity-based sleep monitoring (Actigraphy) | 1 week- 6 months
  The actigraph is a wristwatch-like device attached to the child's wrist, which enables continuous recording of the child's movements for extended periods, with no interference with the child's natural sleep environment.
  The following actigraphic sleep measures will be included in this study: (a) sleep onset time (b) total sleep duration from sleep onset to morning rising time; (c) morning rising time; (d) sleep percentage; (e) true sleep time; and (f) number of night-wakings.

CONTACTS AND LOCATIONS:
Overall Officials: Avi Sadeh, Prof., Study Director — Tel Aviv University; Schneider Children's Medical Center of Israel
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel, Israel